CLINICAL TRIAL: NCT05365386
Title: Evaluation of the Efficacy and Safety of a Thermal Fractional Skin Treatment System (TIXEL®) for the Treatment of Facial and / or Scalp Actinic Keratoses.
Brief Title: Efficacy and Safety of Tixel Treatment on Facial and/or Scalp Actinic Keratoses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novoxel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 0827
Record Dates: First submitted 2022-03-23; First posted 2022-05-09 (Actual); Results first posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Actinic Keratoses
Keywords: actinic keratoses.
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: Single-center, Prospective, Open Label, with Before-After Study Design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tixel Treatment (Experimental): All subjects will undergo 1-3 treatments (determined by the investigator assessment), 3-4 weeks apart with the Tixel device.
  Interventions: Device: Tixel C

INTERVENTIONS:
Device: Tixel C — This is a non-invasive thermo-mechanical treatment to the scalp and/or face using the Tixel technology.

SUMMARY:
Evaluation of the Efficacy and Safety of a thermal fractional skin treatment system (Tixel) for the treatment of facial and/or scalp actinic keratoses

DETAILED DESCRIPTION:
Single-center, Prospective, Open-Label, with Before-After Study Design. Up to 25 subjects will be enrolled to the study to provide at least 20 evaluable subjects. Subjects will be examined to determine the severity and extent of actinic keratoses.

All subjects will undergo 1-3 treatments (determined by the investigator assessment), 3-4 weeks apart.

Follow-up visits will be performed after the last treatment visit: 4 weeks (±7 days) and 12 weeks (±7 days).

The inclusion criteria would be mild to moderate thickness confluent actinic keratoses located to scalp and/or face.

Each subject will participate in the study for up to 20 weeks. Total study duration is estimated to be up to 12 months from enrollment of the first subject until last subject visit (including FUs).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, age 18-80 years old.
2. Skin Phototype I-VI.
3. Subject has mild to moderate thickness confluent AKs on his/her scalp and/or face.
4. Subject is willing and able to comply with protocol requirements and all study visits.
5. Subject has provided written informed consent.

Exclusion Criteria:

1. Any patient who has undergone tanning during the 4 weeks prior to any treatment session and/or any patient who plans to undergo tanning during the 4 weeks following any treatment session (patients who may be exposed to the sun for short periods of time occasionally are not contra-indicated as long as they apply a high SPF sunscreen (>50).
2. Current active Herpes Simplex infection.
3. Current skin cancer, malignant sites and/or advanced premalignant lesions or moles in the treatment area.
4. An impaired immune system condition or use of immunosuppressive medication.
5. Collagen disorders, keloid formation and/or abnormal wound healing.
6. Any patient who takes or has taken any medications (including via topical application), herbal treatment (oral or topic), food supplements or vitamins, which may cause fragile skin or impaired skin healing during the last 3 months.
7. Any patient who has used oral retinoids within 6 months prior to treatment or less.
8. Any patient who has a history of bleeding coagulopathies.
9. Any patient who has tattoos or permanent makeup in the treated area.
10. Any patient who has burned skin, blistered skin, irritated skin, or sensitive skin in any of the areas to be treated.
11. Women who are pregnant (as determined by self-reporting), lactating, or less than 3 months post-delivery, possibly pregnant or planning a pregnancy during the study period.
12. Currently participating in or recently participated in another clinical trial (within the last 30 days).
13. Prior treatment with ablative laser, any laser or photo-dynamic therapy 3 months prior to enrollment.
14. Any cryotherapy or electrodessication 6 weeks prior to enrollment.
15. Systemic retinoid therapy within 6 months prior to enrollment, topical treatment with 5-Fluorouracil cream and/or imiquimod cream and/or diclofenac gel 6 months prior to enrollment.
16. Prior treatment with Tixel.
17. Face cannot be treated due to dermal disorder other than AKs, such as infection, surgical treatment etc.
18. Subject has a systemic disease manifested by AKs (e.g. immune suppression).
19. Significant systemic illness.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Assi Levi, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Ha'Sharon Campus, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tixel Treatment
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: A total of 20 subjects were enrolled in the study. All subjects were included in the PP population. All subjects received the full treatment sessions and had photos from the 12-week FU visit and therefore, completed the study.
Arm/Group | Tixel Treatment
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Israel | 20

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Tixel for Treatment of Actinic Keratosis
Description: The overall mean percentage reduction in actinic keratoses lesion count performed by the investigator manually, confirmed and documented using photograph images taken at baseline and at 12 weeks follow-up visit (or 12-weeks post last treatment if less than 3 treatments were done) (before and after marking the present actinic keratoses using a washable eyeliner) calculated as the relative change from baseline at 12 weeks. New lesions which were not existed in baseline will not be counted.
Time Frame: up to 12 weeks post last treatment
Population: per protocol population - subject lesion count change from baseline % at 12 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Tixel Treatment
Number analyzed (Participants) | 20
percentage change | -90.4 (14.7)

2. Secondary Outcome: Efficacy Evaluation of Tixel for Treatment of Actinic Keratosis
Description: The mean change in actinic keratoses lesion count, performed by the investigator manually, confirmed and documented using photograph images, from baseline at 4 and 12 weeks follow-up visit.
Time Frame: up to 12 weeks post last treatment
Population: per protocol population - subject lesion count change from baseline at 4 and 12 weeks FU
Measure: Mean (Standard Deviation); unit: Number of lesions counted
Arm/Group | Tixel Treatment
Number analyzed (Participants) | 20
Number of lesions counted
  Baseline - Total No. of leasions counted | 10.0 (9.7)
  4 weeks FU - Total No. of lesions counted -Change from Baseline | 8.1 (6.8)
  12 weeks FU - Total No. of lesions counted -Change from Baseline | 8.5 (6.9)

3. Secondary Outcome: Efficacy Evaluation of Tixel for Treatment of Actinic Keratosis
Description: The overall mean percentage reduction in actinic keratoses lesion count performed by the investigator manually, confirmed and documented using photograph images taken at baseline and at 4 weeks follow-up visit (before and after marking the present actinic keratoses using a washable eyeliner) calculated as the relative change from baseline at 4 weeks follow-up visit. New lesions which were not existed in baseline will not be counted.
Time Frame: up to 4 weeks post last treatment
Population: per protocol population - subject lesion count change from baseline % at 4 weeks
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Tixel Treatment
Number analyzed (Participants) | 20
percentage change | -83.6 (16.9)

4. Secondary Outcome: Efficacy of Tixel for Treatment of Actinic Keratosis - Percentage of Subjects That Demonstrated Reduction in Actinic Keratosis Lesion Count 3 Months After the Last Treatment.
Description: * Percentage of subjects that demonstrate a 26-50% in reduction in actinic keratoses lesion count 3 months after the final treatment.
  * Percentage of subjects that demonstrate a 51-75% in reduction in actinic keratoses lesion count 3 months after the final treatment.
  * Percentage of subjects that demonstrate more than 76% in reduction in actinic keratoses lesion count 3 months after the final treatment.
Time Frame: up to 12 weeks post last treatment
Population: Lesion count - relative change from baseline (by category)
Measure: Count of Participants; unit: Participants
Arm/Group | Tixel Treatment
Number analyzed (Participants) | 20
Participants
  0-25% | 0
  26-50% | 1
  51-75% | 1
  76-99% | 8
  100% | 10

5. Secondary Outcome: To Evaluate the Subject's Satisfaction.
Description: Subjects' satisfaction assessed at the final follow-up visit (based on the subject experience questionnaire which includes 3 questions relating to treatment results, treatment experience and treatment expectations) graded on a score of 1- 5; 1 being not satisfied and 5 being very satisfied).
Time Frame: up to 12 weeks post last treatment
Population: per protocol population - Experience questionnaire completed by the subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Tixel Treatment
Number analyzed (Participants) | 20
Participants
  I am satisfied with the results of the treatment (Improvement Assessment): Excellent - Very satisfied (score 5) | 19
  I am satisfied with the results of the treatment (Improvement Assessment): Good - Satisfied (score 4) | 1
  I am satisfied with the results of the treatment (Improvement Assessment): Moderately - satisfied (score 3) | 0
  I am satisfied with the results of the treatment (Improvement Assessment): Fair - Satisfied to some extent (score 2) | 0
  I am satisfied with the results of the treatment (Improvement Assessment): Poor - Poor or not satisfied at all (score 1) | 0
  I am satisfied with the treatment experience: Excellent - Very satisfied (score 5) | 19
  I am satisfied with the treatment experience: Good - Satisfied (score 4) | 1
  I am satisfied with the treatment experience: Moderately - satisfied (score 3) | 0
  I am satisfied with the treatment experience: Fair - Satisfied to some extent (score 2) | 0
  I am satisfied with the treatment experience: Poor - Poor or not satisfied at all (score 1) | 0
  The treatment has fulfilled my expectations: Excellent - Very satisfied (score 5) | 16
  The treatment has fulfilled my expectations: Good - Satisfied (score 4) | 4
  The treatment has fulfilled my expectations: Moderately - satisfied (score 3) | 0
  The treatment has fulfilled my expectations: Fair - Satisfied to some extent (score 2) | 0
  The treatment has fulfilled my expectations: Poor - Poor or not satisfied at all (score 1) | 0

6. Secondary Outcome: Safety Evaluation - Adverse Events
Description: Procedure-related Adverse events during the study.
Time Frame: up to 12 weeks post last treatment
Population: safety population - Procedure-related Adverse Events reported
Measure: Count of Participants; unit: Participants
Arm/Group | Tixel Treatment
Number analyzed (Participants) | 20
Participants | 0

7. Secondary Outcome: Subject Subjective Downtime Assessment
Description: Defined as the period of time following the procedure during which the subject felt unable/unwilling to go out in public due to skin reactions. The assessment will be recorded by the subject using the Subject Subjective Downtime Assessment following each treatment and will be collected at the site at the follow-up visits up to 4 weeks FU following treatment 3 (third treatment).
Time Frame: up to 4 weeks post last treatment
Population: Downtime was assessed at the FU visits post treatments.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Tixel Treatment
Number analyzed (Participants) | 20
Hours
  Follow-Up & Treatment 2. Time until return to work: number analyzed (Participants) | 19
  Follow-Up & Treatment 2. Time until return to work | 1.7 (5.7)
  Follow-Up & Treatment 2. Time until return to Social activities: number analyzed (Participants) | 19
  Follow-Up & Treatment 2. Time until return to Social activities | 1.4 (5.5)
  Follow-Up & Treatment 2. Sensasion of heat: number analyzed (Participants) | 19
  Follow-Up & Treatment 2. Sensasion of heat | 7.8 (19.6)
  Follow-Up & Treatment 2.Redness: number analyzed (Participants) | 19
  Follow-Up & Treatment 2.Redness | 44.3 (48.7)
  Follow-Up & Treatment 2. Edema: number analyzed (Participants) | 19
  Follow-Up & Treatment 2. Edema | 10.7 (22.9)
  Follow-Up & Treatment 2. Scabs: number analyzed (Participants) | 19
  Follow-Up & Treatment 2. Scabs | 40.4 (81.6)
  Follow-Up & Treatment 3. Time until return to work: number analyzed (Participants) | 19
  Follow-Up & Treatment 3. Time until return to work | 1.4 (5.5)
  Follow-Up & Treatment 3. Time until return to Social activities: number analyzed (Participants) | 19
  Follow-Up & Treatment 3. Time until return to Social activities | 4.1 (12.0)
  Follow-Up & Treatment 3. Sensation of heat: number analyzed (Participants) | 19
  Follow-Up & Treatment 3. Sensation of heat | 0.7 (2.8)
  Follow-Up & Treatment 3.Redness: number analyzed (Participants) | 19
  Follow-Up & Treatment 3.Redness | 33.4 (55.2)
  Follow-Up & Treatment 3. Edema: number analyzed (Participants) | 19
  Follow-Up & Treatment 3. Edema | 1.3 (5.5)
  Follow-Up & Treatment 3. Scabs: number analyzed (Participants) | 19
  Follow-Up & Treatment 3. Scabs | 54.2 (93.6)
  4 weeks FU Time until return to work | 0.1 (0.4)
  4 weeks FU Time until return to Social activities | 0.2 (0.7)
  4 weeks FU sensation of heat | 1.5 (5.3)
  4 weeks FU Redness | 36.1 (36.1)
  4 weeks FU Edema | 2.5 (7.4)
  4 weeks FU Scabs | 36.0 (59.0)

8. Secondary Outcome: VAS Assessment
Description: Procedure related pain by the subjects using VAS for pain of 0-10 where a higher score indicates greater pain.
Time Frame: up to 8 weeks (treatments period)
Population: The mean procedure-associated VAS scores reported by the subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tixel Treatment
Number analyzed (Participants) | 20
score on a scale
  mean procedure-associated VAS scores - treatment 1 | 2.0 (2.0)
  mean procedure-associated VAS scores - treatment 2: number analyzed (Participants) | 19
  mean procedure-associated VAS scores - treatment 2 | 1.9 (1.7)
  mean procedure-associated VAS scores - treatment 3: number analyzed (Participants) | 19
  mean procedure-associated VAS scores - treatment 3 | 1.7 (1.7)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the initiation of the treatment until the end of the study period, and a total duration of 12 weeks of FU completion.
Description: Reported adverse events.
Arm/Group | Tixel Treatment
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tixel Treatment (N=20)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-16): https://cdn.clinicaltrials.gov/large-docs/86/NCT05365386/Prot_SAP_000.pdf